CLINICAL TRIAL: NCT03455634
Title: Treatment of Malocclusion Class II/1 - Predictors for Seeking, Compliance and Outcome
Brief Title: Predictors Associated With Seeking Orthodontic Treatment, Compliance and Treatment Success
Acronym: PONCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visnja Katic (Other)
Collaborators: Clinical Hospital Center Rijeka (Other); University of Rijeka (Other)
Responsible Party: Sponsor-Investigator, Visnja Katic, Post-doc, University of Rijeka
Organization: University of Rijeka (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2170-24-01-15-2; 2170-29-02/1-14-5 (Other: Clinical Hospital Center Rijeka, Croatia); 13.06.2.1.53 (Other Grant/Funding Number: University of Rijeka); uniri-biomed-18-22 (Other Grant/Funding Number: University of Rijeka); IP9 (Other Grant/Funding Number: J. J. Strossmayer University of Osijek, Faculy of Dental Medicine and Health)
Record Dates: First submitted 2018-02-21; First posted 2018-03-06 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Malocclusion, Angle Class II
Keywords: quality of life
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Twin Block (Active Comparator): Twin Block functional appliance
  Interventions: Device: Twin Block
- Sander (Active Comparator): Sander bite jumping appliance
  Interventions: Device: Sander bite jumping appliance
- Control (No Intervention): no intervention

INTERVENTIONS:
Device: Twin Block — functional appliances for the stimulation of the mandibular growth
  Arms: Twin Block
Device: Sander bite jumping appliance — functional appliances for the stimulation of the mandibular growth
  Arms: Sander

SUMMARY:
Aim: to search for reasons for seeking orthodontic treatment, compliance during orthodontic treatment, drop-out from orthodontic treatment and success of orthodontic treatment.

Methods: evaluation before, during and at the end of orthodontic treatment. Clinical and diagnostic evaluation of complexity before and at the end of orthodontic treatment, evaluation of awareness of treatment need, impact on social and psychological aspects, functional disturbances, impact of malocclusion on quality of life, social interaction, ability to perform daily activities.

DETAILED DESCRIPTION:
Data will include diagnostic measurements on study casts, x-rays, and data from questionnaires given to children and parents. Statistical analyses will explore predictors of treatment success with treatment need, compliance and psycho-social domains.

ELIGIBILITY:
Inclusion Criteria:

* distal molar occlusion, overjet >5 mm, cervical vertebral maturation method stages (CS) -CS2, CS3 or CS4

Exclusion Criteria:

* mental retardation

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Overjet | baseline
  sagittal distance between upper and lower anterior teeth measured in mm
Child perception questionnaire age 11-14 (CPQ 11-14 SF16) , subscale measuring oral symptoms | baseline
  CPQ 11-14, answers on 5-point Likert scale (0-4), score range 0-16, higher score means greater impact of oral symptoms on quality of life
subscale functional limitations of CPQ 11-14 SF16 | baseline
  CPQ 11-14, answers on 5-point Likert scale (0-4), score range 0-16, higher score means greater impact of functional limitations on quality of life
subscale emotional well-being of CPQ 11-14 SF16 | baseline
  CPQ 11-14, answers on 5-point Likert scale (0-4), score range 0-16, higher score means greater impact of emotional wee-being on quality of life
subscale social well-being of CPQ 11-14 SF 16 | baseline
  CPQ 11-14, answers on 5-point Likert scale (0-4), score range 0-16, higher score means greater impact of social well-being on quality of life
Self-perceived satisfaction with dental appearance | baseline
  rating scale, answer on 5-point Likert scale (0-4), higher score means greater satisfaction with dental apperance
Self-perceived treatment need | baseline
  rating scale, answers on 5-point Likert scale (0-4), higher score means greater self-perceived treatment need
overall score of CPQ 11-14 SF 16 and SF8 | baseline
  CPQ 11-14, answers on 5-point Likert scale (0-4), score range 0-32 for SF8 and 0-64 for SF16 (sum of all items in short-form 8 and 16 instruments), higher score means higher impact of oral disorders on quality of life
change in overjet | change from baseline to one year of appliance wear
  sagittal distance between upper and lower anterior teeth measured in mm

SECONDARY OUTCOMES:
Parental-Caregiver Perceptions Questionnaire (P CPQ), subscale oral symptoms | baseline
  P CPQ, answers on 5-point Likert scale (0-4), score range 0-24, higher score means greater impact of children's oral health status on oral symptoms, as perceived by parents / caregivers
P CPQ, subscale functional limitations | baseline
  P CPQ, answers on 5-point Likert scale (0-4), score range 0-28, higher score means greater impact of children's oral health status on functional limitations, as perceived by parents / caregivers
P CPQ, subscale emotional well-being | baseline
  P CPQ, answers on 5-point Likert scale (0-4), score range 0-32, higher score means greater impact of children's oral health status on emotional well-being, as perceived by parents / caregivers
P CPQ, subscale social well-being | baseline
  P CPQ, answers on 5-point Likert scale (0-4), score range 0-40, higher score means greater impact of children's oral health status on social well-being, as perceived by parents / caregivers
overall score of P CPQ | baseline
  P CPQ, answers on 5-point Likert scale (0-4), score range 0-124 (sum of subscales), higher score means greater impact of children's oral health status on quality of life, as perceived by parents / caregivers
parental/family activity subscale of Family Impact Scale (FIS) questionnaire | baseline
  FIS questionnaire, answers on 5-point Likert scale (0-4), score range 0-20, higher score means greater impact of children's oral health status on parental/family activity, as perceived by parents / caregivers
parental emotions subscale of FIS | baseline
  FIS, answers on 5-point Likert scale (0-4), score range 0-16, higher score means greater impact of children's oral health status on parental emotions, as perceived by parents / caregivers
family conflict subscale of FIS | baseline
  FIS, answers on 5-point Likert scale (0-4), score range 0-16, higher score means greater impact of children's oral health status on family conflict, as perceived by parents / caregivers
financial burden subscale of FIS | baseline
  FIS, answers on 5-point Likert scale (0-4), score range 0-4, higher score means greater impact of children's oral health status on financial burden, as perceived by parents / caregivers
overall score of FIS | baseline
  FIS, answers on 5-point Likert scale (0-4), score range 0-56 (sum of subscales), higher score means greater impact of children's oral health status on family, as perceived by parents / caregivers
change in oral symptoms of CPQ 11-14 SF16 | change from baseline to one year of appliance wear
  CPQ 11-14, answers on 5-point Likert scale (0-4), score range 0-16, change in sum score from baseline to one year of appliance, higher score means greater impact of change of oral symptoms on quality of life
change in functional limitations of CPQ | change from baseline to one year of appliance wear
  CPQ 11-14, answers on 5-point Likert scale (0-4), score range 0-16, change in sum score from baseline to one year of appliance, higher score means greater impact of change in functional limitations on quality of life
change in emotional well-being of CPQ | change from baseline to one year of appliance wear
  CPQ 11-14, answers on 5-point Likert scale (0-4), score range 0-16, change in sum score from baseline to one year of appliance, higher score means greater impact of change in emotional well-being on quality of life
change in social well-being of CPQ | change from baseline to one year of appliance wear
  CPQ 11-14, answers on 5-point Likert scale (0-4), score range 0-16, change in sum score from baseline to one year of appliance, higher score means greater impact of change in social well-being on quality of life
change in overall score of CPQ SF8 | change from baseline to one year of appliance wear
  CPQ 11-14, answers on 5-point Likert scale (0-4), score range 0-32, change in sum score from baseline to one year of appliance, higher score means greater impact of change in oral disorders on quality of life
validation of CPQ 11-14 in Croatia | one year
  16 items and 8 items short form questionnaires, answers on 5-point Likert scale (0-4), score range 0-64, higher score means greater impairment of quality of life
validation of P CPQ in Croatia | one year
  31 items, answers on 5-point Likert scale (0-4), score range 0-124, higher score means greater impairment of childrens' quality of life perceived by their parents
validation of FIS in Croatia | one year
  14 items, answers on 5-point Likert scale (0-4), score range 0-56, higher score means greater impairment of children's' quality of life perceived by their parents

CONTACTS AND LOCATIONS:
Overall Officials: Stjepan Spalj, Study Director — University of Rijeka Faculty of Dental Medicine
Locations (1):
- University of Rijeka, Faculty of Dental Medicine, Rijeka, Primorsko-goranska County, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Brumini M, Slaj M, Katic V, Pavlic A, Trinajstic Zrinski M, Spalj S. Parental influence is the most important predictor of child's orthodontic treatment demand in a preadolescent age. Odontology. 2020 Jan;108(1):109-116. doi: 10.1007/s10266-019-00447-1. Epub 2019 Aug 23. PMID 31444594
- [Result] Acev DP, Brumini M, Slaj M, Katic V, Spalj S. Child Perceptions Questionnaire in Croatia: Two Domains for Measuring Oral Health. Acta Stomatol Croat. 2019 Mar;53(1):47-54. doi: 10.15644/asc53/1/5. PMID 31118532
- [Result] Uhac M, Zibar Belasic T, Perkovic V, Zigante M, Spalj S. Validation of the Parental-Caregivers Perception Questionnaire (P-CPQ) in Croatia. Abstract book 6th Congress of School of Dental Medicine, University of Zagreb. Acta Stomatol Croat. 2020;54:210:212.
- [Result] Brumini M, Uhac M, Zibar Belasic T, Spalj S. Parental attitude and emotional well-being mediate orthodontic treatment demand in adolescents. Abstract book 6th Congress of School of Dental Medicine, University of Zagreb. Acta Stomatol Croat. 2020;54:210:212-3.
- [Result] Brumini M. Predictors of orthodontic treatment demand in early adolescence (dissertation). Rijeka; University of Rijeka, Faculty of Medicine: 2020.
- [Result] Uhac M, Zibar Belasic T, Perkovic V, Matijevic M, Spalj S. Orthodontic treatment demand in young adolescents - Are parents familiar with their children's desires and reasons? Int J Paediatr Dent. 2022 May;32(3):383-391. doi: 10.1111/ipd.12893. Epub 2021 Nov 28. PMID 34402117
- [Result] Uhač M, Zibar Belašić T, Perković V, Matijević M, Špalj S. Orthodontic treatment demand in young adolescents - comparison of parents and their children. 7. Međunarodni kongres Stomatološkog fakulteta Sveučilišta u Zagrebu. Acta Stomatologica Croatica. Rovinj, Hrvatska, 21.-22.05.2021.
- [Result] Spalj S, Uhac M, Brumini M. Role of parents in patient compliance during class II division 1 malocclusion. 51st SIDO International Congress on-line. 13-14.11.2020.
- [Result] Marijanović M, Uhač M, Žigante M, Špalj S. Validation of the Family Impact Scale (FIS) in Croatia. 1. Kongres Fakulteta dentalne medicine u Rijeci. 1. i 2. listopada 2020.
- [Result] Brumini M, Špalj S. Child Perceptions Questionnaire - validation protocol. 8th Virtual world congress of dental students. Zagreb, 20.-22.05.2020.
- [Result] Uhač M, Žigante M, Špalj S. Early Childhood Oral Health Impact Scale and orthodontics: cross-cultural adaptation in Croatia. 51st SIDO International Congress on-line. 13-14.11.2020.
- [Derived] Cukaj Ademi H, Zigante M, Premaraj Thyagaseely S, Tudor V, Palomo JM, Spalj S. Mandibular Advancement in Dentofacial Orthopaedics: Effects on Pharyngeal Airway, Dentoskeletal Characteristics and Quality of Life: A Randomised Controlled Trial. Orthod Craniofac Res. 2026 Feb;29(1):122-133. doi: 10.1111/ocr.70056. Epub 2025 Nov 10. PMID 41211711